CLINICAL TRIAL: NCT03710759
Title: Effect of Assisted Autogenic Drainage In Children Suffering From Pneumonia - a Quasi Experimental Study
Brief Title: Effect of Assisted Autogenic Drainage In Children Suffering From Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC Summyia Siddique
Record Dates: First submitted 2018-10-13; First posted 2018-10-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Pneumonia Childhood
Keywords: Pneumonia; Drainage; Autogenic Drainage
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Assistive Autogenic Drainage (Experimental): Autogenic drainage (AD) is a breathing technique that uses controlled breathing and least amount of coughing to clear secretions from your chest. It involves you hearing and feeling your secretions as you breathe out and controlling the urge to cough until secretions are high up and easily cleared with little effort.
  Interventions: Other: Assistive autogenic Drainage

INTERVENTIONS:
Other: Assistive autogenic Drainage — Assistive autogenic Drainage : All the 3 components of Autogenic drainage was given passively to the patients. By placing the hands on the child's chest, the therapist manually increases the expiratory flow to achieve the different lung volume breathing.

SUMMARY:
Quasi experimental study with duration will be of 6 month, data will be collected from Fauji Foundation Hospital, Rawalpindi. Sample size was calculated from open epi tool (2017) was n=60. Non probability convenient type of sampling technique is used. Children suffering from pneumonia between the ages 5-15 years with class III & IV on pneumonia severity index. Both genders are included under study. Patients on 2nd & 3rd generation anti-biotic therapy for pneumonia are included in the study. Children with musculoskeletal disorders, neuromuscular disorders, cardiovascular co-morbidities and children with diagnosed lobular pneumonia will be excluded. Self-structured questionnaire will be used which includes the demographics, Pneumonia Severity Index, type of Assistive Breathing devices/ Litre of Oxygen support, Vitals, Atrial blood gases(ABG's), Chest X rays and Pediatric Early Warning Sign-Respiratory system.

DETAILED DESCRIPTION:
Pneumonia is the number one infectious killer of children under age 5 globally, according to a World Health Organization (WHO) report year 2015, about 9,35,002 children die of pneumonia every year. In the same report it is stated that Pakistan ranks at third among 15 countries contributing to the global burden of child pneumonia. Pneumonia is basically an infection in one or both lungs. It can be caused by bacteria, viruses, or fungi. Bacterial pneumonia is the most common type in infants however in children Respiratory Syncytial Virus (RSV) is most common cause of Viral Pneumonia. Regarding the pathophysiology of Pneumonia, there is an inflammation in the air sacs of lungs, which are called alveoli, resultantly the alveoli are filled with fluid or pus, making it difficult for the patient to breathe. In order to clear the airways assistive techniques are used besides standard airway management. Autogenic drainage (AD) is an airway clearance technique which utilizes controlled breathing at different lung volumes in order to loosen, mobilize and move secretions in three stages towards the larger central airways.One of the modified form of Autogenic Drainage is Assisted Autogenic Drainage (AAD) which is based upon the principles of Autogenic Drainage and is used in infants and younger patient groups. This technique is performed by placing the hands on the child's chest, the therapist manually increases the expiratory flow in order to achieve the different lung volume breathing.

The chapter 07: vol 1 of book "Physiotherapy Intervention" states that the aim of AAD is to achieve an optimal expiratory flow progressively through all generations of bronchi without causing dynamic airway collapse. In 2007 on " Forced expiratory technique, directed cough and autogenic drainage" and sates that these techniques in combined manner are effective in producing significant results.The direct method of chest percussion was first described by Auenbrugger as reported by the European Respiratory Journal, later it was used globally. The Chochrane Library published a research review on Chest physiotherapy for pneumonia in children in 2012, stating that Autogenic drainage is effective in treating cystic fibrosis (CF). In March 2017 on " The use of assisted autogenic drainage in children with acute and chronic respiratory disease" in population of South Africa which states that AAD is of significance importance while treating chronic respiratory diseases however the efficacy in direct effect on acute respiratory diseases is not studied before.In 1998 conducted a study on the topic of "Alternatives to percussion and postural drainage: A review of mucus clearance therapies: AD, positive expiratory pressure (PEP), Flutter valve, Intrapulmonary percussive ventilation and high frequency with Thira vest." Since late 1990's work has continuously been done on chronic respiratory diseases like Cystic Fibrosis in relation with Autogenic Drainage however regarding Assisted Autogenic Drainage in children suffering from Pneumonia, there is not much work done according to my knowledge. A study conducted in March 2017 in population of South Africa which states that AAD is of significance importance while treating chronic respiratory diseases however the efficacy in direct effect on acute respiratory diseases is not studied before. This study will be going to add Evidence Based Treatment in the practice of Cardiopulmonary Rehabilitation and could be effective treatment of Pneumonia in Children population through Assisted Autogenic Drainage technique of chest clearance. It will be helpful in treating children suffering from Pneumonia by adding literature using an evidence based Chest Physical therapy treatment.

According to the consort guidelines of the assessment of manuscript the only limitation found in the parent study was that the study title included both infants and young children however only infants were actually recruited in the study. The objective of my current study is to determine the effects of Assisted Autogenic Drainage in children with pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* class III & IV on pneumonia severity index.
* Both genders are included under study.
* Patients on 2nd & 3rd generation anti-biotic therapy for pneumonia are included.

Exclusion Criteria:

* Children with Musculoskeletal, Neuromuscular and Cardiovascular co-morbidities.
* Children with diagnosed lobular pneumonia are also excluded.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-05-30 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Atrial Blood Gases | Day 07
  change from baseline Atrial Blood Gases (PH, carbon dioxide partial pressure (PCO2), partial pressure of Oxygen PO2, saturation SPO2)

SECONDARY OUTCOMES:
Pulse rate | Day 1
  change from baseline pulse rate
Pulse rate | Day 3
  change from day 1 pulse rate
Pulse rate | Day 7
  change from day 3 pulse rate
Respiratory | Day 1
  change from baseline Respiratory rate
Respiratory | Day 3
  change from day 1 Respiratory rate
Respiratory | Day 7
  change from day 3 Respiratory rate
Chest Xray | Day 7
  change of chest Xrays From baseline
Pediatric Early Warning System (PEWS) | Day 1
  change of PEWs from baseline
Pediatric Early Warning System (PEWS) | Day 3
  change of PEWs from day 1
Pediatric Early Warning System (PEWS) | Day 7
  change of PEWs from day 3

CONTACTS AND LOCATIONS:
Overall Officials: Sumaiyah Obaid, MSPT, Principal Investigator — Riphah International University
Locations (1):
- Fauji Foundation Hospital, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chisti MJ, Tebruegge M, La Vincente S, Graham SM, Duke T. Pneumonia in severely malnourished children in developing countries - mortality risk, aetiology and validity of WHO clinical signs: a systematic review. Trop Med Int Health. 2009 Oct;14(10):1173-89. doi: 10.1111/j.1365-3156.2009.02364.x. PMID 19772545
- [Background] Alcon A, Fabregas N, Torres A. Pathophysiology of pneumonia. Clin Chest Med. 2005 Mar;26(1):39-46. doi: 10.1016/j.ccm.2004.10.013. PMID 15802164
- [Background] Pryor JA. Physiotherapy for airway clearance in adults. Eur Respir J. 1999 Dec;14(6):1418-24. doi: 10.1183/09031936.99.14614189. PMID 10624775
- [Background] Wallaert E, Perez T, Prevotat A, Reychler G, Wallaert B, Le Rouzic O. The immediate effects of a single autogenic drainage session on ventilatory mechanics in adult subjects with cystic fibrosis. PLoS One. 2018 Mar 29;13(3):e0195154. doi: 10.1371/journal.pone.0195154. eCollection 2018. PMID 29596479
- [Background] Corten L, Jelsma J, Human A, Rahim S, Morrow BM. Assisted autogenic drainage in infants and young children hospitalized with uncomplicated pneumonia, a pilot study. Physiother Res Int. 2018 Jan;23(1). doi: 10.1002/pri.1690. Epub 2017 Jul 19. PMID 28722167
- [Background] Abdelbasset W, Elnegamy T. Effect of chest physical therapy on pediatrics hospitalized with pneumonia. International Journal of Health and Rehabilitation Sciences. 2015;4(4):219-26.
- [Background] Agostini P, Knowles N. Autogenic drainage: the technique, physiological basis and evidence. Physiotherapy. 2007 Jun 1;93(2):157-63.
- [Background] Chaves GS, Fregonezi GA, Dias FA, Ribeiro CT, Guerra RO, Freitas DA, Parreira VF, Mendonca KM. Chest physiotherapy for pneumonia in children. Cochrane Database Syst Rev. 2013 Sep 20;(9):CD010277. doi: 10.1002/14651858.CD010277.pub2. PMID 24057988
- [Background] Akre M, Finkelstein M, Erickson M, Liu M, Vanderbilt L, Billman G. Sensitivity of the pediatric early warning score to identify patient deterioration. Pediatrics. 2010 Apr;125(4):e763-9. doi: 10.1542/peds.2009-0338. Epub 2010 Mar 22. PMID 20308222
- [Background] Monaghan A. Detecting and managing deterioration in children. Paediatr Nurs. 2005 Feb;17(1):32-5. doi: 10.7748/paed2005.02.17.1.32.c964. No abstract available. PMID 15751446
- [Background] Fleming S, Thompson M, Stevens R, Heneghan C, Pluddemann A, Maconochie I, Tarassenko L, Mant D. Normal ranges of heart rate and respiratory rate in children from birth to 18 years of age: a systematic review of observational studies. Lancet. 2011 Mar 19;377(9770):1011-8. doi: 10.1016/S0140-6736(10)62226-X. PMID 21411136
- [Background] Gajdos V, Katsahian S, Beydon N, Abadie V, de Pontual L, Larrar S, Epaud R, Chevallier B, Bailleux S, Mollet-Boudjemline A, Bouyer J, Chevret S, Labrune P. Effectiveness of chest physiotherapy in infants hospitalized with acute bronchiolitis: a multicenter, randomized, controlled trial. PLoS Med. 2010 Sep 28;7(9):e1000345. doi: 10.1371/journal.pmed.1000345. PMID 20927359